CLINICAL TRIAL: NCT02261714
Title: A Phase I/II Trial of TG01 and Gemcitabine as Adjuvant Therapy for Treating Patients With Resected Adenocarcinoma of the Pancreas
Brief Title: Antigen-specific Cancer Immunotherapy (TG01) and Gemcitabine as Adjuvant Therapy in Resected Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Targovax ASA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT TG01-01
Record Dates: First submitted 2014-03-24; First posted 2014-10-10 (Estimated); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer, Resected
Keywords: Pancreatic cancer, resected; Vaccine; KRAS
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TG01/GM-CSF and Gemcitabine (Experimental)
  Interventions: Biological: TG01

INTERVENTIONS:
Biological: TG01 — TG01 and GM-CSF will be administered on days 1, 8, 15, 22 and 36. TG01 alone will also be given on days 36 and 50 for DTH assessment. Gemcitabine will start at least 3 weeks after TG01/GM-CSF and will be given on days 1, 8 and 15 of a four-weeks cycle up to 6 cycles in total.
  Once chemotherapy is completed, GM-CSF and TG01 injections will resume and will be given every 4 weeks from the end of the chemotherapy period up to week 52 (plus once at week 5 post-chemotherapy) and then every 12 weeks from week 52 to week 104. TG01 alone will be given 8 weeks after the end of chemotherapy for DTH assessment.
  TG01 will be given at a dose of 0.70 mg/injection and GM-CSF will be given at a dose of 30 micrograms both as intradermal injections.
  Gemcitabine will be given at a dose of 1000 mg/m2 iv over 30 minutes
Biological: TG01 — For patients not able to start TG01 quickly after surgery, the vaccination can start at the same time as the chemotherapy as long as they start within 12 weeks from surgery. Gemcitabine will start at the same time as TG01/GM-CSF and will be given on days 1, 8 and 15 of a four-weeks cycle up to 6 cycles in total.
  TG01 will be given at a dose of 0.70 mg/injection and GM-CSF will be given at a dose of 30 micrograms both as intradermal injections.
  Gemcitabine will be given at a dose of 1000 mg/m2 iv over 30 minutes

SUMMARY:
The purpose of this study is to investigate the effect of TG01 and Granulocyte macrophage colony stimulating factor (GM-CSF) when given in addition to gemcitabine (chemotherapy) and

* Understand any possible side effects of the additional use of TG01/GM-CSF with gemcitabine
* Investigate whether TG01/GM-CSF when given with gemcitabine can produce an immune response
* Investigate if the treatment can delay or reduce recurrence of the disease

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed diagnosis of adenocarcinoma of the pancreas
2. Stage I or II disease (clinical stage T1-3, N0-1, M0 by AJCC staging criteria).
3. Successful surgical resection

   * Complete resection (R0) or with microscopic residual disease (R1)
   * Expected to receive gemcitabine monotherapy as adjuvant chemotherapy
4. Laboratory Values:

   * Absolute neutrophil count ≥ 1.5 x 10^9/l
   * Platelets ≥100 x 10^9/l
   * Haemoglobin ≥ 9 g/dl
   * Total bilirubin ≤ 1.5 x UNL
   * Serum creatinine ≤ 1.5 x UNL
   * Albumin ≥ 2.5 g/dl
   * AST or ALT ≥ 5 x UNL
5. 18 years of age or older.
6. ECOG performance status (PS) of 0-1.
7. Life expectancy of at least 6 months
8. Men and women of childbearing potential must be willing to use effective methods of contraception to prevent pregnancy
9. Provide written (signed) informed consent to participate in the trial prior to any trial specific screening procedures

Exclusion Criteria:

1. Has received an investigational drug within 4 weeks prior to Trial drug administration
2. Has received previous therapy for pancreatic cancer including radiation or chemotherapy (except for the primary resection or primary neoadjuvant chemotherapy).
3. Is currently receiving any agent with a known effect on the immune system, unless at dose levels that are not immunosuppressive (e.g. Prednisone at 10 mg/day or less or as inhaled steroid at doses used for the treatment of asthma).
4. Has any other serious illnesses or medical conditions such as, but not limited to:

   * Any uncontrolled infection
   * Uncontrolled cardiac failure classification III or IV (NY Heart Association)
   * Uncontrolled systemic and gastro-intestinal inflammatory conditions
   * Bone marrow dysplasia
   * History of auto-immune disease
   * History of adverse reactions to vaccines
5. Known history of positive tests for HIV/AIDS, hepatitis B or C
6. Pregnant or lactating females or have no pregnancy test at baseline (postmenopausal women must have been amenorrhoeic for at least 12 months to be considered of non-childbearing potential).
7. Contraindication to gemcitabine treatment
8. Have had any other malignancies within last 3 years (except for adequately treated carcinoma of the cervix or basal or squamous cell skin cancer)
9. Known malignant brain lesion(s)
10. Are unlikely to start chemotherapy within 12 weeks of surgery (e.g. delayed wound healing, or infection, etc.)
11. Are not expected to complete 6 cycles of chemotherapy
12. Are planned to receive yellow fever or other live (attenuated) vaccines during the course of study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-12; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel PALMER, Principal Investigator — University of Liverpool Molecular and Clinical Cancer Medicine /UCD Duncan Building / Daulby Street / Liverpool; Juan VALLE, Principal Investigator — University of Manchester / The Christie NHS Foundation Trust /Wilmslow Road / Manchester; Svein DUELAND, Principal Investigator — Oslo University Hospital HF / the Norwegian Radium Hospital / Ullernchausseen 70 / Oslo; Yuk Ting MA, Principal Investigator — Queen Elizabeth University Hospital / Edgaston / Birmingham; Emiliano Calvo, Principal Investigator — Centro Integral Oncologico Clara Campal / Hospital HM Universitario Sanchinarro / Madrid
Locations (5):
- Oslo University Hospital HF the Norwegian Radium Hospital, Oslo, Norway
- Centro Integral Oncologico Clara Campal / Hospital HM Universitario Sanchinarro, Madrid, Spain
- United Kingdom (3):
  - Queen Elizabeth University Hospital / Edgaston /, Birmingham
  - University of Liverpool / Molecular and Clinical Cancer Medicine, Liverpool
  - University of Manchester / The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Background] Gjertsen MK, Buanes T, Rosseland AR, Bakka A, Gladhaug I, Soreide O, Eriksen JA, Moller M, Baksaas I, Lothe RA, Saeterdal I, Gaudernack G. Intradermal ras peptide vaccination with granulocyte-macrophage colony-stimulating factor as adjuvant: Clinical and immunological responses in patients with pancreatic adenocarcinoma. Int J Cancer. 2001 May 1;92(3):441-50. doi: 10.1002/ijc.1205. PMID 11291084
- [Background] Weden S, Klemp M, Gladhaug IP, Moller M, Eriksen JA, Gaudernack G, Buanes T. Long-term follow-up of patients with resected pancreatic cancer following vaccination against mutant K-ras. Int J Cancer. 2011 Mar 1;128(5):1120-8. doi: 10.1002/ijc.25449. PMID 20473937
- [Derived] Palmer DH, Valle JW, Ma YT, Faluyi O, Neoptolemos JP, Jensen Gjertsen T, Iversen B, Amund Eriksen J, Moller AS, Aksnes AK, Miller R, Dueland S. TG01/GM-CSF and adjuvant gemcitabine in patients with resected RAS-mutant adenocarcinoma of the pancreas (CT TG01-01): a single-arm, phase 1/2 trial. Br J Cancer. 2020 Mar;122(7):971-977. doi: 10.1038/s41416-020-0752-7. Epub 2020 Feb 17. PMID 32063605

RESULTS

PARTICIPANT FLOW:
Groups:
- TG01/GM-CSF and Gemcitabine: TG01: TG01 and GM-CSF will be administered on days 1, 8, 15, 22 and 36. TG01 alone will also be given on days 36 and 50 for DTH assessment. Gemcitabine will start at least 3 weeks after TG01/GM-CSF and will be given on days 1, 8 and 15 of a four-weeks cycle up to 6 cycles in total. Once chemotherapy is completed, GM-CSF and TG01 injections will resume and will be given every 4 weeks from the end of the chemotherapy period up to week 52 (plus once at week 5 post-chemotherapy) and then every 12 weeks from week 52 to week 104. TG01 alone will be given 8 weeks after the end of chemotherapy for DTH assessment.
  TG01 will be given at a dose of 0.70 mg/injection and GM-CSF will be given at a dose of 30 micrograms both as intradermal injections.
  Gemcitabine will be given at a dose of 1000 mg/m2 iv over 30 minutes TG01: For patients not able to start TG01 quickly after surgery, the vaccination can start at the same time as the chemotherapy as long as they start within 12 weeks from surge
Period: Overall Study
Arm/Group | TG01/GM-CSF and Gemcitabine
Started | 32
Completed | 4
Not Completed | 28

BASELINE CHARACTERISTICS:
Arm/Group | TG01/GM-CSF and Gemcitabine
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 16
Age, Continuous [Mean (Full Range); unit: Years] | 64.1 [46 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 31
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  Norway | 11
  United Kingdom | 21

OUTCOME MEASURES:

1. Primary Outcome: Patients' Safety During Study
Description: Assess the safety (number and nature of Adverse events and laboratory data occurring during study (before, during and after chemotherapy is given) in subjects treated with the Pancreatic Cancer ASCI
Time Frame: 2 years
Measure: Number; unit: Events related to TG01 and /or GM-CSF
Arm/Group | TG01/GM-CSF and Gemcitabine
Number analyzed (Participants) | 32
Events related to TG01 and /or GM-CSF
  AEs related to TG01 and/or GM-CSF | 90
  SAEs related to TG01 and/or GM-CSF | 2

2. Primary Outcome: Patients' Immune Response
Description: Assess the Immune response (DTH responses and Proliferative T-cell responses) up to 2 years of treatment
Time Frame: During the 2 years of treatment
Measure: Number; unit: percentage of patients
Groups:
- TG01/GM-CSF and Gemcitabine: TG01: TG01 and GM-CSF will be administered on days 1, 8, 15, 22 and 36. TG01 alone will also be given on days 36 and 50 for DTH assessment. Gemcitabine will start at least 3 weeks after TG01/GM-CSF and will be given on days 1, 8 and 15 of a four-weeks cycle up to 6 cycles in total. Once chemotherapy is completed, GM-CSF and TG01 injections will resume and will be given every 4 weeks from the end of the chemotherapy period up to week 52 (plus once at week 5 post-chemotherapy) and then every 12 weeks from week 52 to week 104. TG01 alone will be given 8 weeks after the end of chemotherapy for DTH assessment. TG01 will be given at a dose of 0.70 mg/injection and GM-CSF will be given at a dose of 30 micrograms both as intradermal injections. Gemcitabine will be given at a dose of 1000 mg/m2 iv over 30 minutes TG01: For patients not able to start TG01 quickly after surgery, the vaccination can start at the same time as the chemotherapy as long as they start within 12 weeks from surgery.
Arm/Group | TG01/GM-CSF and Gemcitabine
Number analyzed (Participants) | 32
percentage of patients | 94

3. Secondary Outcome: Clinical Efficacy
Description: Efficacy exploring disease free survival and overall survival.
Time Frame: DFS was followed for up to 2 years and OS until last patient included had been in the study for 3 years.
Measure: Median (Full Range); unit: Months
Arm/Group | TG01/GM-CSF and Gemcitabine
Number analyzed (Participants) | 32
Months
  Overall survival | 33.3 [24.0 to 40.0]
  Disease free survival | 16.1 [11.1 to 19.6]

4. Other Pre Specified Outcome: Relationship Between (KRAS) Status and Clinical Efficacy
Description: Relationship between KRAS status and recurrence
Time Frame: 2 years
Population: As the majority of the patients (26 of 32) patients had a KRAS mutation detected, it was not possible to accurately assess relationship between KRAS status and survival outcomes.
Arm/Group | TG01/GM-CSF and Gemcitabine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | TG01/GM-CSF and Gemcitabine
All-Cause Mortality (participants affected / at risk) | 18/32
Serious Adverse Events (participants affected / at risk) | 3/32
Other Adverse Events (participants affected / at risk) | 16/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG01/GM-CSF and Gemcitabine (N=32)
Pyrexia (General disorders) | 1 (2)
Anaphylactic reaction (Immune system disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG01/GM-CSF and Gemcitabine (N=32)
Nausea (Gastrointestinal disorders) | 16 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/14/NCT02261714/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT02261714/SAP_001.pdf